CLINICAL TRIAL: NCT05461820
Title: Clinical Study on the Effect of Routine Treatment and Intensive Treatment on the Regulation of Graves' Disease and the Cumulative Recurrence Two Years After Drug Withdrawal
Brief Title: Effects of Different Treatment Schemes on the Regulation and Recurrence of Graves' Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-SR-037
Record Dates: First submitted 2022-05-04; First posted 2022-07-18 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Graves Disease; Relapse; Treatment; Drug Withdrawal
MeSH Terms: conditions — Graves Disease; Recurrence; Substance Withdrawal Syndrome | interventions — Methimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional treatment group (Active Comparator): According to the thyroid function, if the initial free thyroxine(FT4) ≥ 3 times the normal value, the initial dose of methimazole is 30mg/ day, the thyroid function will be tested every four weeks, and the dose will be reduced when thyroid stimulating hormone(TSH) > normal lower limit or free triiodothyronine(FT3) < normal lower limit or FT4 < normal lower limit. The dose will be reduced according to the clinical routine, specifically, every day (30 mg→20 mg→10 mg→5mg→2.5 mg) If the initial FT4 is less than 3 times the normal value, the initial dose of methimazole is 15mg/ day, and the thyroid function is tested every four weeks. When TSH is greater than the normal lower limit or FT3 is less than the normal lower limit or FT4 is less than the normal lower limit, the dose will be reduced according to the clinical routine, specifically every day for 24 months. If TSH > 100 mIU/L occurs during the treatment, the reduction speed will be accelerated, and 1-2 dose levels can be skipped.
  Interventions: Drug: Methimazole
- Intensive treatment group (Active Comparator): If the initial FT4≥ 3 times of normal value, the initial dose of methimazole was 30mg/ day, and the thyroid function and antibodies were detected every four weeks. When TSH≥4.2 mIU/L, the amount of methimazole began to decrease, specifically in a daily manner (30 mg→20 mg→15mg). The dose was maintained after the decrease to 15 mg. In the case of hypothyroidism, levothyroxine was added until the three antibodies (TPOAb, TGAb and TRAb) were negative. The dose was maintained for six months, and then the doses of methimazole and levothyroxine were gradually reduced until drug discontinuation (each month). If the initial FT4 was less than 3 times of normal level, the initial dose of methimazole was 15 mg/ day, and levothyroxine was added when hypothyroidism occurred. After all three antibodies were negative, the doses were gradually reduced to the point of drug discontinuation.
  Interventions: Drug: Methimazole

INTERVENTIONS:
Drug: Methimazole — Methimazole used in this study was produced by Merck, Germany, and its trade name is Thyrozol. The specification of this drug is 10mg/ tablet, and its validity period is 36 months. It was approved by FDA in 2009 and listed in China in 2011.
  Other Names: Thyrozol

SUMMARY:
In this study, the dose of methimazole was adjusted according to the different states of thyroid function, and the effects of conventional therapy and intensive therapy on the cumulative recurrence of Graves' hyperthyroidism after two years of drug withdrawal were evaluated. At the same time, the changes of immune indexes and inflammatory factors in the regulation process were evaluated. This study is a phase IV clinical study designed and carried out by the First Affiliated Hospital of Nanjing Medical University (Jiangsu Province Hospital), which is a randomized, open and routine treatment group with parallel control.

DETAILED DESCRIPTION:
The results show that the high recurrence rate of antithyroid drugs may be related to the insufficient treatment time, the fact that thyroid autoantibodies did not turn negative when the drugs were stopped, and the thyroid volume did not shrink after treatment. However, individual differences are large, and there is no clear conclusion yet. Graves hyperthyroidism is a common organ-specific autoimmune disease, and its diagnosis mainly depends on the detection of thyroid autoantibodies, especially thyroid-stimulating receptor (TRAb). The antigens in thyroid gland include thyroglobulin (Tg), thyroid peroxidase (TPO) and sodium iodide symporter (NIS) besides thyroid stimulating receptor (TR). Graves hyperthyroidism patients were not only positive for TRAb, but also some patients were positive for anti-thyroglobulin antibody (TgAb) and anti-thyroid peroxidase antibody (TPOAb). At present, the traditional antithyroid drug treatment scheme is to adjust the dosage according to whether the thyroid function returns to normal or not, and observe the antibody turning negative at the same time, and only pay attention to whether TRAb turns negative or not. It has been found that whether TPOAb turns negative when stopping the drug can predict the recurrence after stopping the drug, suggesting that it is not only necessary to observe whether TRAb turns negative, but also to pay attention to whether other thyroid autoantibodies turn negative during the treatment of hyperthyroidism. The negative conversion of all antibodies may indicate that autoantigens are no longer exposed, and the immune balance is stable.

Methimazole (MMI) is one of the most important antithyroid drugs in the treatment of Graves' disease. It mainly blocks the synthesis of thyroid hormone by inhibiting the activity of peroxidase and reduces the production of thyroid hormone. At the same time, some studies have found that methimazole has immunomodulatory effect. Methimazole is recommended for initial treatment of first-time Graves' hyperthyroidism. 30mg/d is suitable for severe Graves' hyperthyroidism and 15mg/d is suitable for mild and moderate Graves' hyperthyroidism. Research has used blocking alternative methods to treat hyperthyroidism patients, maintaining the moderate or high dose of methimazole without decreasing, such as adding levothyroxine to treat hypothyroidism when hypothyroidism occurs, in order to suppress the immune state of Graves' disease patients. However, the research results have not found that it can reduce the recurrence rate of hyperthyroidism. Analyzing the results of these clinical studies, it is found that the use time of methimazole in some studies of blocking replacement therapy is short, and the total treatment time is only one year, and all antibodies are not required to turn negative at the end of treatment. Some studies only focus on the negative conversion of TRAb antibody, but not on the negative conversion of other antibodies such as TgAb and TPOAb.

Therefore, in this study, the intensive treatment group was treated with the inhibition substitution method of fixed middle dose methimazole plus levothyroxine, and the antibody was reduced after all turned negative, while the conventional treatment group was reduced according to whether the thyroid function was normal, so as to evaluate the effects of intensive treatment and conventional treatment on the cumulative recurrence of Graves' hyperthyroidism after two years of drug withdrawal. At the same time, the changes of immune indexes and inflammatory factors during the regulation process were evaluated. To provide evidence for improving the clinical remission rate of Graves' hyperthyroidism and exploring the etiology of Graves' hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Graves hyperthyroidism (responsible for doctors' clinical diagnosis)
* Age 18-65, for both men and women
* Thyroid receptor antibody (TRAb) was positive
* Take part in this research voluntarily and sign the informed consent form

Exclusion Criteria:

* Those who have used glucocorticoid or other immunosuppressants for a long time within 3 months before being selected
* Those who have participated in any other drug trials within 3 months before being selected
* Subjects who are participating in clinical research of other drugs
* Patients with a history of malignant tumors
* Ill-controlled hypertension: diastolic blood pressure≥100mmHg, systolic blood pressure ≥160 mmHg
* Blood routine: the total number of white blood cells < 3.0×109 or neutrophils < 1.5× 109
* Other thyroid diseases: such as subacute thyroiditis, thyroid nodules, high-function adenoma
* Alanine aminotransferase(ALT) or aspartate amino transferase(AST) is greater than 2 times of the normal upper limit; When ALT or AST is less than 2 times of the normal upper limit, and the test of hepatitis B two half-and-half positive
* Renal insufficiency: serum creatinine is higher than the upper limit of normal value
* Patients with heart failure
* Patients with coronary heart disease
* Patients with other autoimmune diseases
* Patients who are known to be allergic to any component of this medicine are allergic to the active ingredients or any auxiliary materials in the prescription
* Patients with multiple drug allergies, allergic diseases, people with high sensitivity and drug addicts
* Alcoholism, mental disorder or other observers who are not suitable for drug testing
* Pregnant and lactating women cannot rule out the possibility of pregnancy
* Taking any medicine with unknown ingredients or using traditional Chinese medicine, the researcher judges the medicine that may affect the curative effect of hyperthyroidism
* According to the researcher's judgment, other medical history that reduces the possibility of joining the group or complicates the joining of the group, such as frequent changes in the working environment, may easily lead to lost follow-up.

Rejection Criteria:

* The compliance of this clinical trial protocol is < 80% or > 120%;
* Those who did not meet the inclusion criteria or the exclusion criteria were found during the experiment;
* Those who can't cooperate, including those who can't complete the whole course of treatment, don't complete the follow-up as planned, and increase or decrease adjuvant drugs at will;
* During the trial, use other drugs that may affect the curative effect of this trial.

Termination of Research Criteria:

* Those who are allergic or intolerant to this drug;
* Adverse reactions or serious adverse events that patients can't tolerate occur;
* Pregnant women of childbearing age in the experiment;
* Other diseases appear during the treatment, and the treatment of accompanying diseases will interfere with the clinical observers of this medicine;
* The researcher thinks it is inappropriate to continue the experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative recurrence rate between conventional treatment group and intensive treatment group after two years of withdrawal. | Up to 2 years after drug withdrawal
  Patients took medicine according to the course of treatment. Relapse occurs when the thyroid function returns to hyperthyroidism within 2 years after the drug is stopped.
Number of patients with no adverse reactions during the treatment of Graves' disease | Within the treatment period (average 2 years)
  The patient completed the methimazole treatment, and there were no adverse reactions that needed to be stopped. Adverse reactions refer to any symptoms, syndromes or diseases that affect patients' health during clinical research and observation, and also include clinically relevant situations found in the laboratory or other diagnostic processes, such as unplanned diagnosis and treatment measures, withdrawal from research, or clinically significant laboratory examination items. Blood routine, liver function, kidney function and adverse reactions will be recorded during the follow-up.

SECONDARY OUTCOMES:
Cumulative recurrence rate of hyperthyroidism in conventional treatment group and intensive treatment group after stopping treatment for one year. | Up to 1 years after drug withdrawal
  Patients took medicine according to the course of treatment. Relapse occurs when the thyroid function returns to hyperthyroidism within 1 years after the drug is stopped.
Effects of routine treatment and intensive treatment on titer and positive rate of thyroid autoantibodies | During treatment(average 2 years) and within 2 years after drug withdrawal
  Thyroid function and related antibodies were detected every 4 ~ 8 weeks, and the positive rate and titers of thyroid autoantibodies (including TPOAb, TGAb and TRAb) were compared.
Effect of conventional therapy and intensive therapy on thyroid volume | During treatment(average 2 years) and within 2 years after drug withdrawal
  The changes of thyroid volume during treatment and withdrawal were compared.
Effects of conventional therapy and intensive therapy on cytokines | During treatment(average 2 years) and within 2 years after drug withdrawal
  The changes of cytokines before and after different treatments were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, Study Chair — The First Affiliated Hospital with Nanjing Medical University; Xuqin Zheng, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No
The medical records of the subjects (research medical records , laboratory sheets, etc.) will be kept intact in the hospital. The project researchers, ethics committee and project funding department will be allowed to consult the medical records of the subjects. Any public report on the results of this study will not disclose the personal identity of the subjects. We will make every effort to protect the privacy of the subjects' personal medical data within the scope permitted by the laws of the People's Republic of China.